CLINICAL TRIAL: NCT05815979
Title: Evaluation of the Effect of Virtual Reality Based Nasogastric Catheter Application Skills on the Knowledge, Skills and Self-Confidence of Graduate Nursing Students
Brief Title: Evaluation of the Effect of Virtual Reality Based Nasogastric Catheter Application Skills on the Knowledge, Skills and Self-Confidence of Graduate Nursing StudentsGraduate Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-03-2023/23
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Advanced Practice Nursing
Keywords: nursing education research; Nursing, Practical; Students, Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician who performs the analysis of the data will not know which group the students are in, so statistics will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group:virtual reality, low-reality simple simulation dummy/model (Experimental): Presentation of the From this point of view, the research was planned as a randomized, control group, experimental study to evaluate the effect of virtual reality-based nasogastric tube application skill on the knowledge, skills and self-confidence of graduate nursing students. glasses and an information meeting will be held for all students in the experimental group, and the working procedure of the virtual reality glasses will be introduced. Afterwards, students will monitor the practice skill at least once using virtual reality glasses. After the completed follow-up, the students will be asked to practice their nasogastric tube application skill on a simple simulation mannequin/model with low reality in the laboratory environment.
  Interventions: Behavioral: virtual reality
- Control Group:low-reality simple simulation dummy/model (No Intervention): Students will be shown the ability to apply a nasogastric tube on a low-reality simple simulation mannequin/model in the laboratory with a demonstration method by the same researcher. Afterwards, students will be asked to practice the skill of applying a nasogastric tube on a simple simulation manikin/model. While practicing on a low simple simulation mannequin/model, students will be evaluated according to the 'Nasogastric Catheter Application Skill Checklist' by a person who works as a nurse and has a graduate education in the field of Nursing Fundamentals, and the application time of the student's nasogastric tube will be recorded. After the application, the students will be asked to fill the 'Nasogastric Catheter Application Skill Knowledge Test' and 'Self-Confidence Evaluation Form'. In addition, students will be required to fill in the Anxiety, Stress, Satisfaction and Motivation Evaluation Form.

INTERVENTIONS:
Behavioral: virtual reality — Presentation of the virtual reality glasses and an information meeting will be held for all students in the experimental group, and the working procedure of the virtual reality glasses will be introduced. Afterwards, students will monitor the practice skill at least once using virtual reality glasses. After the completed follow-up, the students will be asked to practice their nasogastric tube application skill on a simple simulation mannequin/model with low reality in the laboratory environment.
  Arms: Experimental Group:virtual reality, low-reality simple simulation dummy/model

SUMMARY:
It is important to evaluate the nasogastric tube application skill, which is one of the basic skills training of graduate students who are about to step into the nursing profession, using traditional and virtual reality methods. From this point of view, the research was planned as a randomized, control group, experimental study to evaluate the effect of virtual reality-based nasogastric tube application skill on the knowledge, skills and self-confidence of graduate nursing students. The research is planned to be carried out between 1 March 2023 and 30 June 2024 with graduate nursing students continuing their education in Eskişehir Osmangazi University, Faculty of Health Sciences, Department of Nursing. The universe of the research will consist of 150 students studying in the 4th grade of Eskişehir Osmangazi University, Faculty of Health Sciences, Department of Nursing in the 2023-2024 academic year. Since it is aimed to reach the universe in the research, no sample selection will be made. Students who volunteer to participate in the research will be listed, each student will be given a sequence number, and random assignment will be made to groups A and B with the help of a computer program (www.random.org). Then, which of these groups is the experimental group and which one is the control group, it will be decided by drawing lots. Data collection tools of the study; Personal Information Form consisting of 11 questions about socio-demographic characteristics and nasogastric tube application skill, Nasogastric Tube Application Skill Knowledge Test consisting of 20 questions, Nasogastric Tube Application Skill Checklist consisting of 52 procedure steps, Self-Confidence Evaluation Form (Visual Comparison Scale - and Anxiety, Stress, Satisfaction and Motivation Evaluation Form (Visual Comparison Scale - GKO). This research will be carried out in two stages as design and implementation. In the first stage of the research, there are training for reminding nasogastric tube application skills, knowledge test, preparation of skill checklist and measurement tools, implementation of software suitable for virtual reality glasses according to nasogastric tube application procedure steps and integration with glasses. In the second stage of the study, the evaluation of the knowledge, skills and self-confidence of the control and experimental groups with the applied intervention is considered.

DETAILED DESCRIPTION:
According to the Global Sustainable Development Report, the coming years are expected to be the digital revolution, consisting of continuous developments in artificial intelligence, connectivity, digitization of information, virtual reality (VR), machine use, blockchain technology, robotics, quantum computing and synthetic biology. One of the areas that are rapidly affected by these new technologies is the health sector.

Sarıkoç (2016) recommends the inclusion of virtual reality applications in the education curricula in order to increase the quality of the education provided and to adapt to the technological developments of the age in the institutions that provide training to healthcare professionals in our country. The World Health Organization also recommends the use of simulation methods in nursing education and providing the necessary infrastructure for this in the standards it has published regarding education.

Different teaching methods have been used from past to present to gain NGS practice skill, which is one of the nursing skills. With the advancing technology, there has been a transition from traditional teaching methods to innovative teaching methods. Augmented reality (AR) and VR applications, which are innovative approaches in nursing education, are becoming widespread in order to meet the changing expectations of the digital generation born and grown in the age of technology with the developing educational strategies. Chiang et al. (2017) compared the haptic system and the traditional method in the teaching of NGS application in their research and reported that the virtual reality-based haptic system is effective. According to the results of the research, it is recommended to repeat the application with large samples. Augmented reality, which enables us to feel and live the physical environment in the real world in a lively, dynamic and real-time manner with sensory inputs created through the computer, is also among the innovative education methods. In their research, Aebersold et al. (2018), in which they equipped NGS application skills with augmented reality technology and turned it into a mobile application, stated that they provide more effective and permanent learning than the traditional method, thanks to the mobile education they give to the students regardless of the classroom environment. Mobile applications, which are one of the innovative education methods, also facilitate learning. Turaç and Çalışkan (2018), in a randomized controlled study evaluating the effectiveness of the education given by the hypermedia method in teaching nasogastric tube feeding on nursing students (n: 60), concluded that hypermedia has a positive effect on learning. Chang and Lai (2021), in a study in which 60 nursing students' ability to apply nasogastric tube with virtual reality was evaluated, reported that after the VR experience, most students reported that the nursing skill module allowed them to practice repeatedly without the supervision of an instructor. In a randomized controlled study evaluating the effectiveness of an immersive 3D interactive video program on nasogastric tube feeding on 45 nursing students by Chao et al. (2021), it was concluded that nursing students' NG tube feeding knowledge and self-confidence improved by watching immersive 3D interactive video via VIVEPAPER. students who perform NGS application skills within the scope of skill laboratory practices cannot comprehend the skill sufficiently because they do not have the opportunity to practice the process from start to finish on the basic anatomical model. As it can be understood from here, one of the most important problems in nursing education is the difficulty of transforming the theoretical knowledge that the student has into a skill. Among the reasons for this; The high number of students, the low number of instructors, the inability to give every student the opportunity to practice, the time constraint, the lack of appropriate laboratory environments and models reduce the effectiveness of teaching. For this reason, it will be important to increase the quality of education by integrating innovative technologies into laboratory environments. The use of these innovative educational technologies in the world literature is limited in our country. There is a need for more research to evaluate the effectiveness of innovative practices by integrating technology into nursing education and practices, not being indifferent to the rapidly developing technology. For this reason, it is important to evaluate the nasogastric tube application skill, which is one of the basic skills training of graduate students who are about to step into the nursing profession, using traditional and virtual reality methods. From this point of view, the research was planned as a randomized, control group, experimental study to evaluate the effect of virtual reality-based nasogastric tube application skill on the knowledge, skills and self-confidence of graduate nursing students.

Research Hypotheses

H0,1: There is no significant difference between the knowledge test mean scores of the students who received training in virtual reality, traditional method and nasogastric tube application.

H1,1: There is a significant difference between the knowledge test mean scores of the students who received training in virtual reality, traditional method and nasogastric tube application.

H0,2: There is no significant difference between the skill checklist mean scores of the students who received training in virtual reality, traditional method and nasogastric tube application.

H1,2: There is a significant difference between the skill checklist mean scores of the students who received training in virtual reality, traditional method and nasogastric tube application.

H0,3: There is no significant difference between the self-confidence scores of the students who received training in virtual reality, traditional method and nasogastric tube application.

H1,3: There is a significant difference between the self-confidence scores of the students who received training in virtual reality, traditional method and nasogastric tube application.

The research is planned to be carried out between 1 March 2023 and 30 June 2024 with graduate nursing students continuing their education in Eskişehir Osmangazi University, Faculty of Health Sciences, Department of Nursing. The universe of the research will consist of 150 students studying in the 4th grade of Eskişehir Osmangazi University, Faculty of Health Sciences, Department of Nursing in the 2023-2024 academic year. Since it is aimed to reach the universe in the research, no sample selection will be made.

Randomization Students who volunteer to participate in the research will be listed, each student will be given a sequence number and randomly assigned to groups A and B with the help of a computer program (www.random.org). Then, which of these groups is the experimental group and which one is the control group, it will be decided by drawing lots. The co-researcher who performed the randomization has no idea about any student and does not know them. In order to avoid bias in skill assessment, the assessment of students according to the skill checklist will be done by a graduate student in nursing fundamentals who is not in the research, working as a nurse. The statistician who performs the analysis of the data will not know in which group the students received data, thus statistical blinding will be provided.

Data collection tools of the study; Personal Information Form consisting of 11 questions about socio-demographic characteristics and nasogastric tube application skill, Nasogastric Tube Application Skill Knowledge Test consisting of 20 questions, Nasogastric Tube Application Skill Checklist consisting of 52 procedure steps, Self-Confidence Evaluation Form (Visual Comparison Scale - and Anxiety, Stress, Satisfaction and Motivation Evaluation Form (Visual Comparison Scale - GKO).

Application of Research This research will be carried out in two stages as design and implementation. In the first stage of the research, there are training for reminding nasogastric tube application skills, knowledge test, preparation of skill checklist and measurement tools, implementation of software suitable for virtual reality glasses according to nasogastric tube application procedure steps and integration with glasses. In the second stage of the study, the evaluation of the knowledge, skills and self-confidence of the control and experimental groups with the applied intervention is considered.

At the beginning of the research, using virtual reality glasses, nasogastric catheter application skill will be prepared in accordance with the process steps, and the software and hardware processes of the system will be developed under the guidance of Eskişehir Osmangazi University Software Engineering. Project applications (such as TÜBİTAK, BEBKA, BAP) will be made for the research budget. With the video designed with virtual reality glasses, it is aimed to gain the skill with the audio-visual presentation of the process steps of the nasogastric tube application skill and the important points to be considered. In the video design that will be integrated into the Virtual Reality Glasses, the content will be simple, understandable and easy to use.

Nasogastric tube application knowledge and skill training is given to nursing students within the scope of Nursing Fundamentals course in the spring semester of the first year. Within the scope of this research, students who graduated by the researcher during the academic term will be given a reminder training with a power point presentation that will last 2 hours in the classroom environment. Reminder training on nasogastric tube application skill will be prepared by the researcher in accordance with the literature. Care will be taken to ensure that the training is clear, concise and simple, in line with the objectives of nasogastric tube application skills. The content validity of the reminder training will be submitted to the opinion of faculty members who are experts in the field of Nursing Principles. Necessary adjustments will be made in line with the feedback received from the experts.

Afterwards, information will be given about the purpose and content of the research. Students who agree to participate in the study will be asked to fill in an informed consent form and a personal information form. Students will be randomly assigned to the experimental and control groups with the randomization program. With the schedule determined after the determined groups, first the control group and then the students in the experimental group will be included in the application. This will prevent groups from being influenced by each other. After the reminder training, laboratory studies for nasogastric tube application will be carried out in the nursing skills laboratory during the week of the training.

Control Group: Students will be shown the ability to apply a nasogastric tube on a low-reality simple simulation mannequin/model in the laboratory with a demonstration method by the same researcher. Afterwards, students will be asked to practice the skill of applying a nasogastric tube on a simple simulation manikin/model. While practicing on a low simple simulation mannequin/model, students will be evaluated according to the 'Nasogastric Catheter Application Skill Checklist' by a person who works as a nurse and has a graduate education in the field of Nursing Fundamentals, and the application time of the student's nasogastric tube will be recorded. After the application, the students will be asked to fill the 'Nasogastric Catheter Application Skill Knowledge Test' and the 'Self-Confidence Evaluation Form (Visual Comparison Scale - GBL)'. In addition, students will be required to fill in the "Anxiety, Stress, Satisfaction and Motivation Evaluation Form" (Visual Comparison Scale - GKO).

Experimental Group: Virtual reality glasses presentation and information meeting will be held for all students in the experimental group, and the working procedure of the virtual reality glasses will be introduced. Afterwards, students will monitor the practice skill at least once using virtual reality glasses. After the completed follow-up, the students will be asked to practice their nasogastric tube application skill on a simple simulation mannequin/model with low reality in the laboratory environment. While practicing on a low simple simulation mannequin/model, students will be evaluated according to the 'Nasogastric Catheter Application Skill Checklist' by a person who is working as a nurse and has a graduate degree in Nursing Fundamentals (the person evaluating the control group), and the nasogastric tube application time of the student will be recorded. After the application, the students will be asked to fill the 'Nasogastric Catheter Application Skill Knowledge Test' and the 'Self-Confidence Evaluation Form (Visual Comparison Scale - GBL)'. In addition, students will be required to fill in the "Anxiety, Stress, Satisfaction and Motivation Evaluation Form" (Visual Comparison Scale - GKO).

ELIGIBILITY:
Inclusion Criteria:

* To graduate from basic high school education,
* Volunteering to participate in the research,
* Being at school on the days of the research,
* Being a senior nursing student
* To be over the age of 18.

Exclusion Criteria:

* Participating in group work
* The student's willingness to participate in the research and then withdraw from the research
* To fill in the data collection forms of the research incompletely
* Having any obstacle that would prevent answering the survey questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form: | on the 1st day of participation in the study
  In the form developed about students' demographic characteristics and nasogastric tube application skills; students' age, gender, the high school they graduated from, their status of seeing themselves suitable for the nursing profession, their preference for the nursing profession, their academic achievement grade point average, their ability to monitor and apply a nasogastric tube in the Fundamentals of Nursing course, their status of applying a nasogastric tube before or watching a video, and There are 11 questions in total, including their experiences with probing application skills.
Nasogastric Catheter Application Skill Checklist | during practice
  Nasogastric Catheter Application Skills Checklist, which was prepared by the researcher, was created according to the process steps for the application skill within the scope of the course content. In the Nasogastric Catheter Application Skills Checklist, there are 52 steps expected to be performed by the students. In the skill checklist, 2 points are given for each complete step, 1 point for each missing step, and 0 point for each uncompleted step. A minimum of 0 points and a maximum of 104 points can be obtained from the "Nasogastric Catheter Application Skills Checklist". Points from the skill checklist will be converted to a 100 point system. As a result of the evaluation, it will be determined that the students' psychomotor skill performances for the application skill increase as the scores obtained from the nasogastric tube application skill checklist increase.As the scores obtained from the skill list increase, the success towards the skill increases.
Self-Confidence Evaluation Form (Visual Comparison Scale - GKO) | within 10 minutes after practice skill
  The GCS is accepted as a safe, valid and usable measurement tool in repeated measurements. GAQ is a 10 cm long scale that can be used horizontally or vertically, starting with "not at all" and ending with "too much". Self-Confidence Evaluation Forum (Visual Comparison Scale - GCS) will be used to determine students' self-confidence level for their ability to apply a nasogastric tube. Then, with the help of a scale divided into 1/10 divisions of the same length as the scale, the evaluation of the student will be graded as "0: no self-confidence and 10: too much self-confidence".A minimum of 0 and a maximum of 10 points is obtained from the scale. As the score obtained from the scale increases, self-confidence increases.
Nasogastric Catheter Application Skill Knowledge Test | A immediately after application skill
  Nasogastric Catheter Application Skill Knowledge Test" was prepared in line with the objectives of the nasogastric tube application skill course content, which was prepared by the researcher according to the literature. The knowledge test is a test that questions students' knowledge necessary for their ability to apply a nasogastric tube. There are 20 questions on the subject in the knowledge test and the lowest 0 and the highest 100 points can be obtained from the test. Each question is evaluated as 5 points. The questions consist of multiple choice statements with five options.As the scores obtained from the knowledge test increase, the success towards the skill increases.
Anxiety, Stress, Satisfaction and Motivation Evaluation Form (Visual Comparison Scale - GKO) | within 10 minutes after practice skill
  The GCS is accepted as a safe, valid and usable measurement tool in repeated measurements. GAQ is a 10 cm long scale that can be used horizontally or vertically, starting with "not at all" and ending with "too much". The Anxiety, Stress, Satisfaction and Motivation Evaluation Forum (Visual Comparison Scale - GCS) will be used to determine the level of anxiety, stress, satisfaction and motivation for students' ability to apply a nasogastric tube. A minimum of 0 and a maximum of 10 points is obtained from the scale.As the score obtained from the scale increases, anxiety, stress, satisfaction and motivation increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Islamic Science and Technology University, Gaziantep, Şahinbey/Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi KS, He X, Chiang VC, Deng Z. A virtual reality based simulator for learning nasogastric tube placement. Comput Biol Med. 2015 Feb;57:103-15. doi: 10.1016/j.compbiomed.2014.12.006. Epub 2014 Dec 17. PMID 25546468
- [Background] Chang YM, Lai CL. Exploring the experiences of nursing students in using immersive virtual reality to learn nursing skills. Nurse Educ Today. 2021 Feb;97:104670. doi: 10.1016/j.nedt.2020.104670. Epub 2020 Nov 17. PMID 33264739
- [Background] Berndt J, Dinndorf-Hogenson G, Herheim R, Hoover C, Lanc N, Neuwirth J, Tollefson B. Collaborative Classroom Simulation (CCS): An Innovative Pedagogy Using Simulation in Nursing Education. Nurs Educ Perspect. 2015 Nov-Dec;36(6):401-2. doi: 10.5480/14-1420. PMID 26753303
- [Background] Vaughn J, Lister M, Shaw RJ. Piloting Augmented Reality Technology to Enhance Realism in Clinical Simulation. Comput Inform Nurs. 2016 Sep;34(9):402-5. doi: 10.1097/CIN.0000000000000251. PMID 27258807
- [Background] Ferguson C, Davidson PM, Scott PJ, Jackson D, Hickman LD. Augmented reality, virtual reality and gaming: an integral part of nursing. Contemp Nurse. 2015;51(1):1-4. doi: 10.1080/10376178.2015.1130360. Epub 2016 Jan 14. No abstract available. PMID 26678947
- [Background] Chao YC, Hu SH, Chiu HY, Huang PH, Tsai HT, Chuang YH. The effects of an immersive 3d interactive video program on improving student nurses' nursing skill competence: A randomized controlled trial study. Nurse Educ Today. 2021 Aug;103:104979. doi: 10.1016/j.nedt.2021.104979. Epub 2021 May 18. PMID 34049120
- [Background] Bankhead R, Boullata J, Brantley S, Corkins M, Guenter P, Krenitsky J, Lyman B, Metheny NA, Mueller C, Robbins S, Wessel J; A.S.P.E.N. Board of Directors. Enteral nutrition practice recommendations. JPEN J Parenter Enteral Nutr. 2009 Mar-Apr;33(2):122-67. doi: 10.1177/0148607108330314. Epub 2009 Jan 26. No abstract available. PMID 19171692
- [Background] Perry, AG. (2016). Enteral Nutrition. In: Elkin, MK., Perry, AG., Potter, PA. (Eds.) Nursing Interventions and clinical skills., Mosby Inc.,St. Louis, Missouri, 996-1036.